CLINICAL TRIAL: NCT05331404
Title: Longitudinal Evaluation of Hearing Aids Rehabilitation Within Age-related Hearing Loss Population : Behavioral and Neuroimaging PET Evaluations.
Brief Title: Evaluation of Hearing Aids Rehabilitation Within Age-related Hearing Loss Population.
Acronym: AGEHEAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/20/0365; 2021-A01993-38 (Other: ID-RCB)
Record Dates: First submitted 2022-04-11; First posted 2022-04-15 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Hearing Loss
Keywords: Presbycusis; Auditory cortex.; Auditory plasticity.; Localization; Speech-in-noise; PET
MeSH Terms: conditions — Hearing Loss; Presbycusis

STUDY DESIGN:
Intervention Model Description: Patient and control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Presbycusis (Experimental): Patients with presbycusis who receive rehabilitation with hearing aids
  Interventions: Radiation: PET examination; Other: Quality of life assessment
- Aged control group (Active Comparator): Aged control group: 15 subjects with normal or near-normal hearing thresholds
  Interventions: Other: Quality of life assessment
- Young control group (Active Comparator): Young control group: 15 subjects with normal hearing thresholds
  Interventions: Radiation: PET examination; Other: Quality of life assessment

INTERVENTIONS:
Radiation: PET examination — PET examinations with auditory stimuli such as human voice and environmental sounds.
  Arms: Presbycusis; Young control group
Other: Quality of life assessment — quality of life assessment by :
  * Speech, Spatial and Qualities of Hearing
  * Hearing Handicap Inventory For The Elderly Screening
  * Short Form Health Survey

SUMMARY:
Hearing aids restore efficiently some auditory functions in age-related hearing loss (ARHL or presbycusis) providing to the elderly an access to oral communication and a return to social life. However, a most of the assessments of their efficacy focus on speech recognition. Spatial hearing and localization are anothers important auditory functions merely evaluated.

The purpose of this study is to evaluate the hearing aids benefits for spatial hearing.

DETAILED DESCRIPTION:
The main objective is to evaluate the hearing aids benefits for spatial hearing with a multidisciplinary approach combing psychophysics, and Positron Emission Tomography (PET) brain imaging in a before/after experimental design. The novelty of the proposal is both theoretical and methodological: the team aim is to identify neural correlates of spatial hearing after hearing rehabilitation and evaluate the evolution of spatial hearing abilities once subjects with presbycusis are fitted with hearing aids. The assessment of spatial hearing processing will rely on both a virtual visuo-auditory 3D immersive platform and functional neuroimaging using PET scan. This project will provide crucial elements for understanding and improving the rehabilitation of age-related hearing loss.

ELIGIBILITY:
Inclusion Criteria:

For presbyacusics subjects:

* Subjects aged over 50 with a difference in symmetrical audiometric thresholds (< 15 dB) between the two ears and requiring hearing aids
* Affiliation to a social security scheme or equivalent
* Acceptance of the protocol and signature of the consent form

For older people with normal hearing:

* Subjects matched in age (+/- 2 years) and gender with the presbycusis group
* Affiliation to a social security scheme or equivalent
* Acceptance of the protocol and signature of the consent form
* Subjects with normal hearing, with hearing thresholds of 20 dB < 2kHz and 40 dB < 4kHz

For young people with normal hearing:

* Subjects aged between 18 and 40 years old,
* Symmetric normal hearing
* Affiliation to a social security scheme or equivalent
* Normally hearing subjects with audiometric thresholds < 20 dB
* Acceptance of the protocol and signature of the consent form

Exclusion Criteria:

* Persons under a legal protection regime for adults (safeguard of justice, guardianship, curator ship, institutionalized, or under mandate for future protection)
* History of associated neurological pathology
* Contraindications to PET
* Cognitive impairment confirmed by the Montreal Cognitive Assessment (MOCA) test (for presbyacusic subjects and normal-hearing elderly subjects)
* Taking psychotropic drugs
* History of epilepsy
* Pregnant or breastfeeding woman
* Participation in another intervention protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
level of brain activity | Month 12
  level of brain activity (in ml/100g/min) measured in the auditory regions in PET when the subject performs a spatial localization task

SECONDARY OUTCOMES:
Life quality by Speech, Spatial and Qualities of Hearing (12) | Month 12
  Speech, Spatial and Qualities of Hearing is a questionnaire specific to the quality of hearing. It has 3 sections; speech hearing, spatial hearing and quality of hearing. This questionnaire contains 15 items evaluated on a scale to 0 (not at all) to 10 (perfectly).
Life quality by Speech, Spatial and Qualities of Hearing (6) | Month 6
  Speech, Spatial and Qualities of Hearing is a questionnaire specific to the quality of hearing. It has 3 sections; speech hearing, spatial hearing and quality of hearing. This questionnaire contains 15 items evaluated on a scale to 0 (not at all) to 10 (perfectly).
life quality by Hearing Handicap Inventory For The Elderly Screening (12) | Month 12
  Hearing Handicap Inventory For The Elderly Screening contains 10 items to identify the social and emotional difficulties encountered by the subject due to his deafness according to specific situations. It makes it possible to detect the handicap perceived by the person (the higher the score, the greater the perception of the handicap due to hearing loss).
life quality by Hearing Handicap Inventory For The Elderly Screening (6) | Month 6
  Hearing Handicap Inventory For The Elderly Screening contains 10 items to identify the social and emotional difficulties encountered by the subject due to his deafness according to specific situations. It makes it possible to detect the handicap perceived by the person (the higher the score, the greater the perception of the handicap due to hearing loss).
life quality by Short Form Health Survey (12) | Month 12
  Short Form Health Survey assesses a patient's overall quality of life. It consists of 36 items.
life quality by Short Form Health Survey (6) | Month 6
  Short Form Health Survey assesses a patient's overall quality of life. It consists of 36 items.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu MARX, Professor, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strelnikov K, Rouger J, Demonet JF, Lagleyre S, Fraysse B, Deguine O, Barone P. Visual activity predicts auditory recovery from deafness after adult cochlear implantation. Brain. 2013 Dec;136(Pt 12):3682-95. doi: 10.1093/brain/awt274. Epub 2013 Oct 17. PMID 24136826
- [Background] Vannson N, James C, Fraysse B, Strelnikov K, Barone P, Deguine O, Marx M. Quality of life and auditory performance in adults with asymmetric hearing loss. Audiol Neurootol. 2015;20 Suppl 1:38-43. doi: 10.1159/000380746. Epub 2015 May 19. PMID 25997394
- [Background] Vannson N, James CJ, Fraysse B, Lescure B, Strelnikov K, Deguine O, Barone P, Marx M. Speech-in-noise perception in unilateral hearing loss: Relation to pure-tone thresholds and brainstem plasticity. Neuropsychologia. 2017 Jul 28;102:135-143. doi: 10.1016/j.neuropsychologia.2017.06.013. Epub 2017 Jun 13. PMID 28623107